CLINICAL TRIAL: NCT00796276
Title: Disposition of Paliperidone Enantiomers After Treatment With Different Formulations of the Racemate and the Separate Enantiomers and the Determination of the Absolute Bioavailability of IR and ER OROS Paliperidone
Brief Title: A Study of Paliperidone Enantiomer Disposition With Different Formulations and the Bioavailability of Immediate- and Extended-release Paliperidone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR004216
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mood disorders; Antipsychotics; Pharmacokinetics; Enantiomer; IR OROS Paliperidone; ER OROS Paliperidone
MeSH Terms: conditions — Schizophrenia; Mood Disorders

INTERVENTIONS:
Drug: IR OROS paliperidone and ER OROS paliperidone

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics of paliperidone in plasma and urine after intravenous (i.v.) administration of the racemate, administration of the immediate-release (IR) racemate oral solution, administration of the ER OROS tablet, and administration of the oral solutions of the individual enantiomers R078543 (+) and R078544 (-); to determine the absolute oral bioavailability of IR and ER OROS paliperidone; to document the (+) and (-) paliperidone enantiomer ratio after i.v. and oral administration (IR and ER OROS paliperidone); to document the possible interconversion between the (+) and (-) enantiomers of paliperidone after oral treatment with the separate enantiomers; to document the possible relationship between the subject's CYP2D6 phenotype and the (+) and (-) enantiomer disposition of paliperidone (CYP2D6 genotyping was used to corroborate the phenotype). In addition, the safety and tolerability of all treatments will be evaluated.

DETAILED DESCRIPTION:
This is a single-center, single-dose, open-label, randomized, crossover study in healthy adults, following a 5-sequence, 5-treatment, 5-period Latin square design. The study consists of a screening phase (within 21 days before the first administration of study drug), and a treatment phase consisting of 5 periods during which volunteers will receive a single dose of study drug under fasting conditions [orally with 240 mL of water or intravenously (i.v.)] in a random order. Pharmacokinetic blood and urine samples will be collected over a 96-hour period following study drug administration during each treatment period. Volunteers will be confined to the testing facility from at least 10 hours before dosing until 72 hours after dosing in each treatment period and will return for additional assessments. Each administration of study drug will be separated by a washout period of at least 7 to a maximum of 14 days. The duration of volunteer participation is maximally 12 weeks, including the 3 week screening period. CYP2D6 metabolizer status will be assessed by phenotyping and will be corroborated by genotyping of a DNA sample to be collected from volunteers who consent to this part of the study. Pharmacokinetic data are available after oral administration of immediate release and extended release formulations of paliperidone. No data are available after i.v. administration of paliperidone. The data obtained in this study for the i.v. route are important to further characterize the pharmacokinetics of paliperidone, and for future population pharmacokinetics modeling of paliperidone. For chiral substances, it is requested by regulatory authority guidelines to document the disposition of the enantiomers. Therefore, the disposition of the (+) and (-) enantiomers of paliperidone for different administration routes (i.v. and oral) and formulations (immediate release and extended release [ER OROS]) will be documented. Separate enantiomers will be administered in this study, as it is important for the full understanding of the pharmacokinetics of paliperidone to document the possible chiral interconversion. Safety and tolerability will be monitored throughout the study. 5 single doses, one each of: Treatment A, 1 mg IR paliperidone oral solution; Treatment B, 3 mg ER OROS paliperidone oral; Treatment C, 1 mg paliperidone as a 30-min i.v. infusion; Treatment D, 1 mg (+)-paliperidone (R078543) oral solution; and Treatment E, 1 mg (-)-paliperidone (R078544) oral solution.

ELIGIBILITY:
Inclusion Criteria:

* Known dextromethorphan (i.e., previously determined) metabolic ratio of <0.02 or >0.35, as determined according to the standard procedures of the study center
* Acceptable weight as defined by body mass index (weight [kg]/height [m²]) range of 18 to 28 kg/m², inclusive
* Normotensive with supine (5 minutes) blood pressure between the range of 100 to 140 mmHg systolic, inclusive, and 60 to 90 mmHg diastolic, inclusive
* Nonsmoking or habitually smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes of tobacco per day for at least 6 months prior to study enrollment
* Healthy on the basis of prestudy screening physical examination, medical history, ECG, and the laboratory results of blood biochemistry, hematology, and urinalysis performed within 21 days before the first study drug dose. If the results of the biochemistry, hematology, or urinalysis testing are not within the reference laboratory ranges, the volunteer can be included only if the investigator judges that the deviations are not clinically significant. For renal function tests, the values must be within the normal laboratory reference ranges
* Women must be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double barrier method, contraceptive transdermal patch, male partner sterilization, and at the discretion of the investigator, total abstinence), postmenopausal for at least 1 year, or surgically sterile before entry and throughout the study
* Women volunteers must also have a negative serum pregnancy test at screening.

Exclusion Criteria:

* Known allergy or history of significant hypersensitivity to heparin, in case a heparin lock will be used
* Drug allergy to risperidone, paliperidone, or any of its excipients
* Recent history of alcohol or substance abuse and/or testing positive for a urine drug screen at study screening
* Relevant history of any cardiovascular, respiratory, neuropsychiatric, renal, hepatic, gastrointestinal (including surgeries, malabsorption problems, or a history of any severe preexisting gastrointestinal narrowing [pathologic or iatrogenic]), endocrine, immunologic diseases, or significant findings on the physical examination
* History of any cancer, with the exception of basal cell carcinoma
* At screening, sustained drops in systolic (>20 mmHg) or diastolic (>10 mmHg) blood pressure after standing for at least 2 minutes which are not associated with an increase in pulse rate of >15 beats per minute
* Positive result for any of the serology tests (hepatitis BsAg, CAb, and HIV-1)
* Consuming more than 450 mg of caffeine per day. This equals 5 cups of tea, 3 cups of coffee, or 8 cans of cola

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-05; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
To characterize and document the pharmacokinetics of paliperidone in plasma and urine;the (+) and (-) paliperidone ratio;the possible interconversion between the (+)- and (-)- enantiomers of paliperidone;the absolute oral bioavailability of paliperidone

SECONDARY OUTCOMES:
To document the possible relationship between the volunteer's CYP2D6 phenotype and the disposition of the (+) and (-) enantiomers of paliperidone and to evaluate the safety and tolerability of the treatments in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of paliperidone enantiomer disposition with different formulations and the bioavailability of immediate- and extended-release paliperidone — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=569&filename=CR004216_CSR.pdf